CLINICAL TRIAL: NCT01445197
Title: A Multicentre, Interventional, Non-randomized, Open-label, Single-group Phase III Study to Evaluate Plasma-Derived Antihaemophilic Factor/Von Willebrand Factor Concentrate (Biostate®) for Immune Tolerance Induction in Male Paediatric Subjects With Haemophilia A (≤ 2%) Who Have Developed High-titre Antibodies to Factor VIII (Factor VIII Inhibitors)
Brief Title: Study of Biostate for Treatment of Children With Hemophilia A Complicated by Antibody Development
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSLCT-BIO-10-67; 2010-020113-85 (EudraCT Number)
Record Dates: First submitted 2011-09-30; First posted 2011-10-03 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-10

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

ARMS (1):
- Biostate (Experimental)
  Interventions: Biological: Biostate

INTERVENTIONS:
Biological: Biostate — 200 IU/kg administered daily

SUMMARY:
This is a clinical study to investigate how well Biostate works in treatment of male patients below the age of 12 years who have a clotting factor deficiency that is aggravated by the development of antibodies. The antibodies are directed against the clotting factor that is given for replacement therapy and usually make therapy unsuccessful. The treatment used in this study is called immune tolerance therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects diagnosed with haemophilia A (≤ 2% FVIII level in the absence of factor replacement, according to their medical history).
* Age 28 days to <12 years.
* Subject is eligible for immune tolerance induction (ITI) therapy

Exclusion Criteria:

* The subject has received ITI previously.
* Subjects with a historical peak inhibitor titre of ≥ 200 BU/mL.
* Concomitant treatment with drugs with immunosuppressive side effects (eg, systemic corticosteroids), azathioprine, cyclophosphamide, high dose immunoglobulin or the use of a protein A column or plasmapheresis and interferons.
* High risk of cardiovascular, cerebrovascular, or other thromboembolic events (excluding catheter thrombosis) as judged by the investigator.
* Subjects who are human immunodeficiency virus (HIV)-1 or HIV-2 positive (as reported in the medical records or determined at screening).

Ages: 28 Days to 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Response to immune tolerance induction (ITI) treatment | 30 months
  Number of subjects who achieve complete, partial, and no response (ITI failure) to treatment.

SECONDARY OUTCOMES:
FVIII inhibitor titre | Up to 65 months
Time to complete response (success) | Up to 65 months
Time to inhibitor titer <0.6 BU/mL for the first time | Up to 65 months
Thromboembolic complications | Up to 65 months
  Number of patients with clinical symptoms or increased markers of coagulation activation
Frequency of bleeding events | Up to 65 months
Number of bleeding events per patient | Up to 65 months
Severity of bleeding events per patient | Up to 65 months
Catheter-related complications | Up to 65 months
  Number of line infections

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Escuriola-Ettingshausen, Principal Investigator — Haemophilia Centre Rhein Main, Frankfurt - Mörfelden
Locations (7):
- Study Site, Vienna, Austria
- Germany (2):
  - Study Site, Frankfurt
  - Study Site, Hamburg
- Greece (2):
  - Study Site, Athens
  - Study Site, Thessaloniki
- Study Site, Milan, Italy
- Study Site, Barnaul, Russia